CLINICAL TRIAL: NCT02694393
Title: Phase I/II Study of Inhaled Sodium Nitrite as an Antimicrobial for Pseudomonas Infection in Cystic Fibrosis
Brief Title: Inhaled Sodium Nitrite as an Antimicrobial for Cystic Fibrosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Protocol closed due to difficulty recruiting subjects and then expiration of investigational product and lack of a manufacturer.
Sponsor: Schmidhofer, Mark, MD (Individual)
Collaborators: Mast Therapeutics, Inc. (Industry); Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Joseph Pilewski, Associate Professor of Medicine and Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO15040062
Record Dates: First submitted 2016-01-11; First posted 2016-02-29 (Estimated); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sodium nitrite (Experimental): Inhalation of 46 or 80 mg of sodium nitrite twice daily for four weeks
  Interventions: Drug: sodium nitrite

INTERVENTIONS:
Drug: sodium nitrite — inhalation of 46 or 80 mg of sodium nitrite by electronic nebulization
  Other Names: AIR001

SUMMARY:
This study will assess the safety of inhaled sodium nitrite in adults with Cystic Fibrosis and chronic Pseudomonas infections, and determine the ability of sodium nitrite to reduce the burden of Pseudomonas.

DETAILED DESCRIPTION:
Pseudomonas aeruginosa infects the airways of 80% of adults with Cystic Fibrosis (CF). In these patients, P. aeruginosa forms extremely antibiotic resistant biofilm communities that accelerate progression of obstructive lung disease. Current treatment of airway infection focuses on monthly cycles of inhaled antibiotics. However up to 20% of adults are infected with multi drug resistant P. aeruginosa for which we have no effective inhaled treatments. These isolates are more common as patients age so with the increasing life expectancy of the CF population, MDR P. aeruginosa is likely to remain a clinical problem. Another 10% of patients are infected with other Gram-negative organisms such as Burkholderia cepacia and Achromobacter species, for which we have inadequate suppressive treatment. Following lung transplant, MDR airway infections remain a problem as the allografts are colonized by strains carried in the paranasal sinuses. Sodium nitrite may present a new antimicrobial approach to treating respiratory infection with Gram-negative organisms, because it is able to prevent biotic biofilm formation.

Within the CF lung, P. aeruginosa grows as a biotic biofilm in association with airway epithelial cells and mucous plaques. This environment has an acidic pH and low oxygen tension with many bacteria subsisting through denitrification (both conditions where traditional antibiotics are less effective). Because biotic biofilms can be up to 500-fold more resistant than biofilms grown on abiotic surfaces, with support from our CF Research Development Program (RDP) Cores, we showed that nitrite prevents biofilm formation on the surface of primary CF airway epithelial cells. Moreover, nitrite dose-dependently potentiates the effects of colistin sulfate in liquid culture, and in biotic biofilms on airway epithelial cells. These data support the hypothesis that nebulized sodium nitrite will inhibit growth of Pseudomonas aeruginosa in CF airways, and identify a potential therapeutic benefit for nitrite alone and cooperatively with colistin as a novel therapy to inhibit P. aeruginosa in CF airways. Nebulized nitrite has been through extensive animal toxicology, and is well tolerated by subjects with pulmonary arterial hypertension where it is being studied as a pulmonary vasodilator.

To determine the therapeutic potential of sodium nitrite for CF, we propose two specific aims:

Aim 1: Determine the safety of nebulized sodium nitrite administered in two doses to patients with CF.

Aim 2: Explore the effects of inhaled sodium nitrite on measures of lung function, exhaled airway nitric oxide, and bacterial burden as measured by quantitative sputum cultures.

To accomplish these aims, we propose a Phase I/II open-label study of sodium nitrite in CF. Key inclusion criteria include individuals over the age 18 with cystic fibrosis as documented by clinical features of CF, and genotyping or a positive sweat test. Exclusion criteria include advanced lung disease, inability to discontinue inhaled antibiotics for four weeks, hospitalization or medication change within 4 weeks of enrollment, baseline systemic hypotension (SBP<90 mm hg), chronic kidney disease (Cr >2.5), severe anemia (Hgb <9 gm/dL in the last six months). The primary outcome is safety, defined as FEV1 measured before and after initial doses on days 0 and 7, and at week 4. Other safety data for the initial doses include pulse oximetry and transcutaneous methemoglobin levels. Secondary endpoints include quantitative sputum cultures, exhaled nitric oxide, sputum nitrite concentration, and patient symptoms as assessed by a CF specific respiratory questionnaire.

Completion of this study will guide the development of sodium nitrite as a single agent for CF infections, and inform future studies examining the effects of sodium nitrite in combination with inhaled colistin for patients with drug resistant bacterial pathogens that are an increasing problem. In addition, the study will provide important safety and efficacy data that may inform future development of inhaled sodium nitrite as a therapy in young patients to augment airway host defense and prevent biofilm formation.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis as documented by clinical features, and documentation of a positive sweat test or two disease causing mutation of the CF gene.

Exclusion Criteria:

* use of supplemental oxygen, FEV1 < 40% predicted, inability to discontinue inhaled antibiotics for 4 weeks,
* hospitalization within 4 weeks prior to enrollment,
* change in maintenance CF therapies within 4 weeks of enrollment,
* severe anemia, significant chronic liver disease, severe pulmonary hypertension, prior organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02; Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pilewski, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Comprehensive Lung Center - Falk Clinic, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Major TA, Panmanee W, Mortensen JE, Gray LD, Hoglen N, Hassett DJ. Sodium nitrite-mediated killing of the major cystic fibrosis pathogens Pseudomonas aeruginosa, Staphylococcus aureus, and Burkholderia cepacia under anaerobic planktonic and biofilm conditions. Antimicrob Agents Chemother. 2010 Nov;54(11):4671-7. doi: 10.1128/AAC.00379-10. Epub 2010 Aug 9. PMID 20696868
- [Background] Zemke AC, Shiva S, Burns JL, Moskowitz SM, Pilewski JM, Gladwin MT, Bomberger JM. Nitrite modulates bacterial antibiotic susceptibility and biofilm formation in association with airway epithelial cells. Free Radic Biol Med. 2014 Dec;77:307-16. doi: 10.1016/j.freeradbiomed.2014.08.011. Epub 2014 Sep 16. PMID 25229185

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had a 2 week wash-out period during which inhaled antibiotics were held before the drug was dosed. If participants had a drop in percent predicted FEV1 between the screening visit and Visit 1 where the drug was dosed, they were excluded from the study. Of our 4 enrolled subjects, 1 subject withdrew from study participation during the washout period and 1 subject failed the wash-out period and was excluded from the study before being assigned to treatment arm.
Groups:
- Nebulized Nitrite: Nebulized nitrite, 40-80 mg
Period: Overall Study
Arm/Group | Nebulized Nitrite
Started | 2
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 25.5 [20 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
FEV1 (Percent predicted) [Mean (Full Range); unit: Percent predicted FEV1] | 61.5 [48 to 75]
exhaled Nitric Oxide [Mean (Full Range); unit: Parts per billion] | 6.5 [5 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Function
Description: forced expiratory volume in one second (FEV1) after inhalation will assess safety
Time Frame: Day 7
Measure: Mean (Full Range); unit: percentage of predicted FEV1
Groups:
- Nebulized Nitrite: Nebulized sodium nitrite, 40-80 mg
Arm/Group | Nebulized Nitrite
Number analyzed (Participants) | 2
percentage of predicted FEV1 | 59 [37 to 81]

2. Primary Outcome: Pulmonary Function
Description: forced expiratory volume in one second (FEV1) after inhalation will assess safety
Time Frame: Day 28
Measure: Number; unit: percentage of predicted FEV1
Arm/Group | Nebulized Nitrite
Number analyzed (Participants) | 1
percentage of predicted FEV1 | 78

3. Secondary Outcome: Exhaled Nitric Oxide
Description: concentration of nitric oxide in exhaled breath
Time Frame: Day 7
Measure: Mean (Full Range); unit: parts per billion
Arm/Group | Nebulized Nitrite
Number analyzed (Participants) | 2
parts per billion | 10 [8 to 12]

4. Secondary Outcome: Exhaled Nitric Oxide
Description: concentration of nitric oxide in exhaled breath
Time Frame: Day 28
Measure: Number; unit: parts per billion
Arm/Group | Nebulized Nitrite
Number analyzed (Participants) | 1
parts per billion | 12

5. Secondary Outcome: Sputum Nitrite Concentration
Description: concentration of nitrite in sputum
Time Frame: day 7
Population: Sputum nitrite data not collected/measured
Arm/Group | Nebulized Nitrite
Number analyzed (Participants) | 0

6. Secondary Outcome: Sputum Nitrite Concentration
Description: concentration of nitrite in sputum
Time Frame: day 28
Population: Sputum nitrite data not collected/measured
Arm/Group | Nebulized Nitrite
Number analyzed (Participants) | 0

7. Secondary Outcome: Pseudomonas Density in Sputum
Description: density of Pseudomonas in sputum
Time Frame: day 28
Population: Pseudomonas density in sputum data not collected/measured
Arm/Group | Nebulized Nitrite
Number analyzed (Participants) | 0

8. Secondary Outcome: CF Questionnaire - Respiratory
Description: respiratory symptom questionnaire
Time Frame: day 28
Population: respiratory symptom questionnaire data not collected/measured
Arm/Group | Nebulized Nitrite
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 42 days following first drug administration visit
Description: The adverse events predicted to be of interest were: methemoglobinemia, hypotension and bronchoconstriction (as measured by FEV1)
Groups:
- Nebulized Nitrite: 40-80 mg nebulized nitrite administration
Arm/Group | Nebulized Nitrite
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebulized Nitrite (N=2)
Methemoglobinemia (Blood and lymphatic system disorders) | 0 (0) — Increase in methemoglobin level measured noninvasively
Hypotension (Cardiac disorders) | 1 (1) — Asymptomatic hypotension in the setting of phlebotomy, resolved without intervention
Decreased FEV1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) — FEV1 decrease of <15% at second

LIMITATIONS AND CAVEATS:
The study was terminated early due to expiration of investigational product and lack of a manufacturer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT02694393/Prot_SAP_000.pdf
  • Informed Consent Form (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02694393/ICF_001.pdf